CLINICAL TRIAL: NCT01294878
Title: Explorative Study on the Use of Omalizumab in Patients Suffering From Interstitial Cystitis/Painful Bladder Syndrome
Brief Title: Omalizumab in Interstitial Cystitis/Bladder Pain Syndrome
Acronym: IComaliz
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: DANIELE PORRU MD, Divisione Urologia, Fondazione IRCCS Policlinico San Matteo, Viale Golgi 19, Pavia 27100, Italy
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: omalizumab-ic
Record Dates: First submitted 2011-02-11; First posted 2011-02-14 (Estimated); Last update posted 2011-02-14 (Estimated); Status verified 2010-12

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome
Keywords: anti-IgE treatment; interstitial cystitis/bladder pain syndrome; omalizumab
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- treatment with omalizumab (Experimental): Treatment was administered subcutaneously every 2 or 4 weeks (according to the calculated total dose) for a total of 48 weeks. Each vial contained 150 mg of the active compound, therefore the number of injections for each administration varied between 1 and 3, depending on the total dose used
  Interventions: Drug: omalizumab

INTERVENTIONS:
Drug: omalizumab — The omalizumab dose has been calculated on the basis of body weight and basal levels of total serum IgE. Treatment was administered subcutaneously every 2 or 4 weeks (according to the calculated total dose) for a total of 48 weeks. Each vial contained 150 mg of the active compound, therefore the number of injections for each administration varied between 1 and 3, depending on the total dose used.
  Other Names: Xolair

SUMMARY:
By hypothesising that Interstitial Cystitis is an allergic disorder of the urogenital system that is linked to mast-cells, current therapy with omalizumab may represent a potential non symptomatic strategy for the treatment of IC/BPS

DETAILED DESCRIPTION:
Interstitial cystitis/Bladder Pain Syndrome is a chronic inflammatory disease of the bladder, that is characterized by pain in the pelvic region and a frequent need to urinate. So far there is not a an effective treatment for this uncommon distressing condition.

The objective of this preliminary study was to evaluate the efficacy of omalizumab in the treatment of Interstitial Cystitis/Bladder Pain Syndrome, evaluated by visual analogue score (VAS) for pain and urgency- frequency, O'Leary-Sant IC symptom and problem index questionnaire (primary outcome), PUF questionnaire and Patient Global Assessment questionnaire, and urination diary (secondary outcomes).

Three female adult patients (24-34 years) suffering form Interstitial Cystitis and chronic bladder pain were included in the study. The omalizumab dose has been calculated on the basis of body weight and basal levels of total serum IgE. Treatment was administered subcutaneously every 2 or 4 weeks (according to the calculated total dose) for a total of 48 weeks. Each vial contained 150 mg of the active compound, therefore the number of injections for each administration varied between 1 and 3, depending on the total dose used. Patients were allowed to take drugs used for IC (Fibrase, Pelvilen, Normast, Quercetin, Chondroitin, Glucosamine per os). During the screening process, the dosage of these drugs was established and stably maintained during the 4 week run-in period.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years, with a range in body weight of 20 and 150 kg, who have provided written informed consent
* In patients diagnosed with IC/PBS that underwent treatment, basal levels of total serum IgE were 30 and 700 IU/ml and patients showed a positive allergic anamnesis (asthma, rhinitis, atopic dermatitis, etc.)
* Diagnosis of IC/PBS was performed according to the criteria established by the National Institute of Health Consensus Conference and patients had symptoms for at least 3 months. Cytoscopy was performed according to the clinical indications

Exclusion Criteria:

* Pregnancy, breastfeeding. Fertile women that did not use secure contraceptive methods (hormonal or double barrier method). Hysterectomized or surgically sterilized women (tubal ligation) and menopause women were admitted into the study.
* Clinically relevant medical conditions (neoplasia, infections, hematologic, renal, hepatic, cardiovascular, hormonal or gastrointestinal pathologies) within 3 months prior to the study. Other specific criteria included patients with positive anamnesis for bladder cancer or affected by actinic cystitis, vaginitis, symptomatic bladder or urethral diverticulum, active genital herpes, bladder or urethral lithiasis.
* Urination frequency less than 5 times per day.
* Known hypersensitivity to any omalizumab component, excipients included (such as monoclonal antibodies, polyclonal gamma globulins)
* Alcohol or drug abuse.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2009-03; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
visual analogue score (VAS) for pain and urgency- frequency | 12 months
  subjective measurement of pain and urgency

SECONDARY OUTCOMES:
PUF questionnaire | 12 months
  assessment of bladder pain and urinary frequency

CONTACTS AND LOCATIONS:
Overall Officials: Daniele Porru, MD, Principal Investigator — Divisione Urologia, Fondazione IRCCS Policlinico San Matteo, Pavia, Italy
Locations (1):
- Divisione Urologia IRCCS Policlinico San Matteo, Pavia, Italy